CLINICAL TRIAL: NCT06902246
Title: Regorafenib and Yttrium-90 Radioembolization for Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Regorafenib and Yttrium-90 Radioembolization for Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Lynn Feun, MD, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230806
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Unresectable Hepatocellular Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Regorafenib in combination with Radioembolization Group (Experimental): Participants in this group will receive combination therapy of Regorafenib and Yttrium 90 Trans-Arterial Radioembolization (Y90 TARE). Participants will receive therapy until unacceptable toxicity, disease progression, or withdrawal of consent, whichever occurs first.
  Total participation duration is approximately 37 months.
  Interventions: Drug: Regorafenib; Radiation: TheraSphere™ Yttrium-90 Trans-Arterial Radioembolization

INTERVENTIONS:
Drug: Regorafenib — Participants will orally self-administer Regorafenib tablets for the first 21 days of each 28-day cycle as follows. Dose-escalation will occur only if there are no significant drug-related adverse events:
  * Safety Run-in Phase: For the first six (6) participants enrolled. The starting dose is 80 mg/day during Cycles 1 and 2. In Cycle 3, the starting dose is 80 mg/day on Days 1 to 7, escalating to 120 mg/day on Days 8 to 14, and then escalating to a maximum dose of 160 mg/day on Days 15 to 21. Participants will continue to receive the maximum tolerated dose determined at the end of Cycle 3.
  * Phase 2: For participants enrolled after the Safety Run-in phase. In Cycle 1, the starting dose is 80 mg/day on Days 1 to 7, escalating to 120 mg/day on Days 8 to 14, and then escalating to a maximum dose 160 mg/day on Days 15 to 21. From Cycle 2 onward, participants will take 160 mg/day (or maximum tolerated dose from Cycle 1), on Days 1 to 21.
  Other Names: Stivarga
Radiation: TheraSphere™ Yttrium-90 Trans-Arterial Radioembolization — Y-90 absorbed glass microspheres will be administered standard of care once via the percutaneous trans-arterial approach after the first 3 weeks of Regorafenib treatment but before Day 28. Additional Y-90 absorbed glass microsphere administration is allowed for treatment of baseline disease in the absence of disease progression within 6 months of the initial Y-90 TARE treatment.
  Other Names: Y-90 TARE

SUMMARY:
The purpose of this study is to determine the effects that Regorafenib in combination with Yttrium-90 (Y-90) radioembolization has on patients with unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ages 18 years old and above.
2. Unresectable Hepatocellular Carcinoma (HCC).
3. Child-Pugh A-B7.
4. Serum bilirubin < 1.5 upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN.
5. Serum creatinine ≤ 1.5 x ULN.
6. International normalized ratio (INR)/Partial thromboplastin time (PTT) ≤ 1.5 x ULN. Note: Participants who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists.
7. Platelet count > 100,000 platelets/mm3, hemoglobin (Hb) 9 g/dL, and absolute neutrophil count (ANC) 1,500 neutrophils/mm3.
8. Mapping angiogram procedure shows radioembolization is feasible and safe to perform.
9. No prior systemic therapy for HCC.
10. Participant agrees to comply with the contraception requirements as described in protocol.

Exclusion Criteria:

1. Angiogram shows vascular shunting which prevents radioembolization.
2. Prior radioembolization.
3. Major extrahepatic disease.
4. Participants with brain metastases.
5. Participants who have not recovered from major surgery. Participants must not undergo any major surgery at or within 30 days prior to study enrollment.
6. Presence of a non-healing wound, non-healing ulcer, or bone fracture.
7. Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
8. Ongoing infection > Grade 2 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
9. Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg [NCI CTCAE v5.0] on repeated measurement) despite optimal medical management.
10. Active or clinically significant cardiac disease including:

    1. Congestive heart failure - New York Heart Association (NYHA) > Class II.
    2. Active coronary artery disease.
    3. Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
    4. Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before study enrollment, or myocardial infarction within 6 months before study enrollment.
11. Evidence or history of bleeding diathesis or coagulopathy.
12. Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
13. Participants with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment or within 6 months of informed consent.
14. Participants with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated ductal carcinoma in situ of the breast, curatively treated nonmelanoma skin carcinoma, noninvasive aerodigestive neoplasms, or superficial bladder tumor. Participants surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before registration are allowed. All cancer treatments must be completed at least 3 years prior to registration.
15. Participants with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2031-01-05 (Estimated); Study Completion 2031-01-05 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) Measured by Number of Participants | Up to 24 months
  Disease Control Rate (DCR) is defined as the number of participants experiencing a best response of complete response (CR), partial response (PR), or stable disease (SD) after receiving protocol therapy. Response will be assessed using modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria for hepatocellular carcinoma.
Number of Participants Experiencing Treatment Related Adverse Events | Up to 25 months
  The number of participants experiencing treatment-related adverse events (AEs) in participants receiving protocol therapy will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5, per physician discretion.
Number of Participants Experiencing Treatment Related Serious Adverse Events | Up to 25 months
  The number of participants experiencing treatment-related serious adverse events (SAEs) in participants receiving protocol therapy will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5, per physician discretion.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  Objective response rate (ORR) is the proportion of patients achieving complete response (CR) or partial response (PR) as the best response. Response will be assessed using modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria for hepatocellular carcinoma.
Time to Tumor Progression | Up to 36 months
  Time-to-tumor progression is defined as the period of time in months from start date of study treatment until documented date of confirmed disease progression. For participants without progression, follow-up time will be censored at the date of last disease assessment (as per mRECIST).
Duration of Overall Response (DOR) | Up to 36 months
  The duration of overall response (DOR) is measured in months from the time measurement criteria are met for complete response (CR) or partial response (PR) per mRECIST criteria, until the first date that recurrent or progressive disease is documented. For participants without progression, follow-up time will be censored at the date of last disease assessment, per mRECIST criteria.
Progression-Free Survival (PFS) | Up to 36 months
  Progression-free survival (PFS) is defined as the elapsed time in months from the first date of study treatment until documented disease progression, per mRECIST criteria or death from any cause, whichever is earlier. For participants who remain alive without progression, follow-up time will be censored at the date of last disease assessment, per mRECIST criteria.
Overall Survival (OS) | Up to 36 months
  Overall survival (OS) is defined as the elapsed time in months from date of first study treatment until death from any cause. Participants without documented death will be censored at the last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn G Feun, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No